CLINICAL TRIAL: NCT00379678
Title: A Pilot Ex-vivo Study to Evaluate the Effect of Pimecrolimus on Antimicrobial Peptide Expression and Vaccinia Virus Growth in Perilesional Skin Cultures of Patients With Atopic Dermatitis
Brief Title: Effects of Pimecrolimus on Skin Biopsy Ex-plants From Patients With Atopic Dermatitis
Status: Completed | Type: Observational
Sponsor: National Jewish Health (Other)
Other Study IDs: HS-2042; Novartis study #CASM981CUS39
Record Dates: First submitted 2006-09-20; First posted 2006-09-22 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- Information not available

SUMMARY:
THe study seeks to determine if pimecrolimus has a positive effect on increasing antimicrobial peptide expression and reducing vaccinia virus growth in the skin explants from patients with atopic dermatitis.

DETAILED DESCRIPTION:
AMP play an important role in the innate immune response against infections. Two major classes of AMP have been identified: the beta defensins (HBD) (Harder 1997) and cathelicidins (LL-37) (Gallo 2002). AMP have been shown to have antibacterial activities against S. aureus (Ong 2002) and antiviral activity against vaccinia virus (VV) (Howell 2004).

The skin of AD patients is characterized by a deficiency in AMP, which may account for their propensity to skin infections (Ong 2002). This AMP deficiency is believed to be due to an increase in Th2 cytokines, IL-4 and IL-13, expression (Ong 2002), as well as an increase of IL-10 expression (Howell 2005). Other cytokines known to affect AMP expression are TNF-alpha (TNFa), IL-6, IL-1 and interferon-gamma (IFN-g). These cytokines induce the expression of AMP (Erdag 2002, Liu 2002, Ong 2002, Nomura 2003). However, negligible levels of TNF-a and IFN-g have been shown in AD skin possibly due to their downregulation by Th2 cytokines (Nomura 2003). Therefore, the neutralization of IL-4, IL-13 and IL-10 in AD patients may correct the AMP deficiency of AD patients and decrease their propensity to recurrent skin infections. Interestingly, the addition of anti-IL10 to skin explants from AD patients augmented HBD-2 and LL-37 expression (Howell 2005). In addition, IL-4 and IL-13 were found to enhance VV replication and down-regulate LL-37 in VV-stimulated keratinocytes and neutralization of IL-4/IL-13 in AD skin augmented LL-37 and inhibited VV replication (Howell 2006a). LL-37 and HBD-3 have been found to kill VV(Howell 2004; Howell 2006b). Thus a deficiency of these AMP may contribute to increased propensity to viral infection. Therapeutic strategies are needed to augment AMP expression in AD skin to reduce skin infection.

Pimecrolimus is a calcineurin inhibitor that binds with high affinity to macrophilin-12. The complex pimecrolimus-macrophilin inhibits calcineurin, a phosphatase required for the dephosphorylation of the cytosolic form of the nuclear factor of activated T cells (NF-AT). As a consequence, pimecrolimus prevents the nuclear translocation of NFAT and thereby the transcription and release of both Th1 and Th2 cytokines such as IL-2, IFN-g, IL-4, IL-5, IL-10, TNF-a and GM-CSF (Grassberger 1999).

As the most common topical corticosteroid treatment used by AD patients, triamcinolone diacetate is included in this study as an active comparator.

ELIGIBILITY:
Inclusion Criteria:

* Has signed the informed consent form
* Male or female of any race and ethnicity
* Patient is 18 years of age or older with active AD
* Active AD of any severity will be defined according to Hanifin and Rajka clinical criteria (Hanifin, J.M., Rajka, G. 1980)
* Chronic AD for more than one year duration

Exclusion Criteria:

* Patients with only AD of the face
* Women of childbearing potential not using the contraception method(s) specified in this study (abstinence, oral contraceptives, IUD,diaphragm), as well as women who are breastfeeding
* Patients with severe medical condition(s) that in the view of the investigator prohibits participation in the study
* Use of any other investigational agent in the last 30 days
* Patient who is pregnant or lactating
* Patient using oral corticosteroids, or any systemic immunosuppressive, or immunomodulary medication within the last 28 days
* Patient who has received immunotherapy within the last year
* Patient with a history of bleeding disorders
* Use of aspirin, oral antihistamines, oral antibiotics, oral cyclosporine, or topical medications within seven days of the Screening/Baseline Visit including (but not restricted to), Elidel, Protopic, topical corticosteroids, and topical antibiotics
* Patients with known lidocaine allergy
* Inability of patient to follow study procedures or documented history of the patient being noncompliant
* Any concomitant diagnosis that, in the opinion of the investigator, might impact the biopsy procedure
* Infected AD
* Use of any topical medication < 7 days or systemic medication < one month prior to study start

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2006-09; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Information not available | Information not available

CONTACTS AND LOCATIONS:
Overall Officials: Donald Leung, MD,PhD, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Medical and Research Center, Denver, Colorado, United States